CLINICAL TRIAL: NCT03744104
Title: Immunogenicity and Safety of a Quadrivalent Influenza Vaccine in Participants Aged Above 3 Years
Brief Title: A Clinical Trial of A Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT060
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadrivalent influenza vaccine (Experimental): Quadrivalent influenza vaccine(containing 2 subtypes of B lineage)
  Interventions: Biological: Quadrivalent influenza vaccine
- Trivalent influenza vaccine A (Active Comparator): Trivalent influenza vaccine (containing B/Victoria lineage)
  Interventions: Biological: Trivalent influenza vaccine A
- Trivalent influenza vaccine B (Active Comparator): Trivalent influenza vaccine (containing B/Yamagata lineage)
  Interventions: Biological: Trivalent influenza vaccine B

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — 0.5 mL, intramuscular, one dose
  Arms: Quadrivalent influenza vaccine
Biological: Trivalent influenza vaccine A — 0.5 mL, intramuscular, one dose
  Arms: Trivalent influenza vaccine A
Biological: Trivalent influenza vaccine B — 0.5 mL, intramuscular, one dose
  Arms: Trivalent influenza vaccine B

SUMMARY:
The aim of this study is to assess the immunogenicity and safety of a quadrivalent influenza vaccine compared with a trivalent influenza vaccine in participants aged above 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of three years,healthy population
* Subjects/ (and the guardian) informed consent, voluntarily participated and signed the informed consent form, with the ability to use thermometers, scales and to fill in diary cards as required
* To comply with the requirements of clinical trial program
* Temperature≤37.0℃ on day of enrollment

Exclusion Criteria:

* A history of influenza virus infection or suspected infection Abnormal blood routine, blood biochemistry and urine routine examination indexes in last three months
* Any prior administration of influenza vaccine in last six months
* Allergy to any component in the vaccine, especially for egg allergy
* Allergy history of any previous vaccination or drug
* Acute episodes of chronic illness or acute illness on the day of vaccination
* Received a live vaccine within fourteen days prior to receiving the vaccine, or received a subunit or inactivated vaccine within seven days
* Congenital or acquired immune deficiencies, or treatment with immunosuppressive agents, such as long-term treatment with systemic corticosteroids
* Suffering from severe chronic diseases (such as Down's syndrome, diabetes, sicklemia or neurological disorders, Green's Barre syndrome)
* Asthma, required urgent treatment in last two years
* The blood products were received prior to the acceptance of the vaccine
* Known or suspected of respiratory disease, acute infection or chronic disease active period, HIV infection, cardiovascular disease, severe hypertension, malignant tumor during treatment, skin diseases
* History of epilepsy, convulsions, or a family history of psychosis
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities), or obvious bruising or coagulopathy
* Plan to move or leave the area for an extended period of time before the end of the study
* Under anti-tb treatment
* Any prior administration of other research medicine/vaccine in last one month
* Women are pregnant or in the near future planned pregnancy or pregnancy test positive

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2688 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Number of participants that presented seroconversion post injection | 30 days after inoculation
  * Seroconvertion is defined as: prevaccination Hemagglutination-inhibition test (HI) antibody titer ≤1:10 and postvaccination HI antibody titer ≥1:40, or prevaccination HI antibody titer ≥1:10 and a postvaccination increase by a factor of four or more.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing
Geometric mean of Hemagglutination-inhibition titre post first study injection | 30 days after inoculation
  * Geometric mean of Hemagglutination-inhibition test titre will be calculated for the different groups of participants post first study injection.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing.

SECONDARY OUTCOMES:
Number of participants that presented seroprotection post injection | 30 days after inoculation
  * Seroprotection is defined as postvaccination Hemagglutination-inhibition test (HI) antibody titer ≥ 1:40.
  * Participants will be collected blood post first study injection, when blood samples will be taken for HI testing
Number of Subjects Reporting Solicited and Unsolicited Adverse Events (AEs) | Continuous observation for 30 days after two inoculations
  * For each group the incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * For each group the incidence rate of subjects with unsolicited AE(s) with 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Hu Yuemei, PhD, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (2):
- China (2):
  - Suining County Center for Disease Control and Prevention, Xuzhou, Jiangsu
  - Xinyi County Center for Disease Control and Prevention, Xuzhou, Jiangsu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03744104/Prot_SAP_000.pdf